CLINICAL TRIAL: NCT03000647
Title: Assessment of the Effectiveness of Guided by a Physiotherapist Versus Non-guided Pelvic Floor Exercises for Urinary Incontinence (UI) in Patients With Relapsing-Remitting (RR) Multiple Sclerosis
Brief Title: Guided Versus Non-guided Pelvic Floor Exercises for Urinary Incontinence in Relapsing-Remitting Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC 65-15 HGV
Record Dates: First submitted 2016-12-14; First posted 2016-12-22 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2018-03

CONDITIONS: Relapsing-Remitting Multiple Sclerosis; Urinary Incontinence
Keywords: Pelvic floor muscle exercise; Supervision; Physiotherapy
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Guided Pelvic floor exercises (Active Comparator): Pelvic floor exercises guided by a physiotherapist
  Interventions: Procedure: Pelvic floor exercises guided by a physiotherapist
- Non-guided pelvic floor exercises (Active Comparator): Pelvic floor exercises not guided
  Interventions: Procedure: Non guided pelvic floor exercises

INTERVENTIONS:
Procedure: Pelvic floor exercises guided by a physiotherapist — Subjects perform two types of contractions of the pelvic floor in two different positions 3 times a day and once a week they check it with a physiotherapist (this day only they do it twice at home)
  Arms: Guided Pelvic floor exercises
Procedure: Non guided pelvic floor exercises — Subjects perform two types of contractions of the pelvic floor in two different positions 3 times a day. They do not attend to meetings with a physiotherapist
  Arms: Non-guided pelvic floor exercises

SUMMARY:
The aim of the study is to evaluate the effectiveness of guided versus non guided pelvic floor exercises for urinary incontinence in patients with Relapsing-Remitting Multiple Sclerosis

DETAILED DESCRIPTION:
Subjects of the study should conduct a specific training in pelvic floor exercises. They were randomly assigned into 2 groups: Group A only received written instructions for exercises to be performed at home; Group B received written instructions and, in addition, exercises were performed in a 30 minutes weekly session with a physiotherapist guiding them

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Relapsing-Remitting Multiple Sclerosis
2. Diagnosed with Urinary Incontinence
3. Minimental Sate Examination (MMSE) scale: More than 24
4. Expanded Disability Status Scale (EDSS) scale: Bladder function 0-4; EDSS 0-6,5
5. Willing to participate in the study
6. Having Signed an informed consent

Exclusion Criteria:

1. Diagnosed with another neurological disease
2. Diagnosed with kidney diseases
3. Having a Relapse of the disease in the last 6 months
4. In Women: Pregnancy os postpartum < 6 months
5. Having gone through surgery for urinary incontinence or prolapses or prostate diseases
6. Having gone through other treatment for pelvic floor
7. MMSE scale: Under 24
8. EDSS scale: Bladder function 5-6 or not knowing; EDSS 7-10
9. ICIQ-SF scale: Severity 19-21
10. Not willing to participate or sign the informed consent form or not able to understand the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Decrease in the number of urinary leakages from baseline | 12 weeks
  Difference in the mean number of leakages (Registered for 3 days with a bladder diary)

SECONDARY OUTCOMES:
Decrease of urinary incontinence severity from baseline | 4,8 and 12 weeks
  Comparison of the results: Questions 1, 2 and 3 of the International Consultation on Incontinence Questionnaire (ICIQ-SF) between the group 1 and 2
Change in quality of life from baseline | 4,8 and 12 weeks
  Comparison of the results (Question 3 of the questionnaire ICIQ-SF and second part (13 questions) of the Overactive Bladder questionnaire (OABQ-SF) between the group 1 and 2
Decrease in the number of urinary leakages from baseline | 4 and 8 weeks
  Comparison of the results (Registered for 3 days with a bladder diary) between the group 1 and 2
Lower urinary tract symptoms from baseline | 4,8 and 12 weeks
  Comparison of de results (First part (6 questions) of the questionnaire OABQ-SF) between the group 1 and 2
Adherence | 12 weeks
  Comparison of the results (Registered with exercise diary)between the group 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Denise Cuevas, BSc, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Hospital General de Villalba, Villalba, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quarto G, Autorino R, Gallo A, De Sio M, D'Armiento M, Perdona S, Damiano R. Quality of life in women with multiple sclerosis and overactive bladder syndrome. Int Urogynecol J Pelvic Floor Dysfunct. 2007 Feb;18(2):189-94. doi: 10.1007/s00192-006-0131-9. Epub 2006 May 13. PMID 16699915
- [Background] Gilpin SA, Gilpin CJ, Dixon JS, Gosling JA, Kirby RS. The effect of age on the autonomic innervation of the urinary bladder. Br J Urol. 1986 Aug;58(4):378-81. doi: 10.1111/j.1464-410x.1986.tb09089.x. PMID 3756405
- [Background] Lucio AC, Campos RM, Perissinotto MC, Miyaoka R, Damasceno BP, D'ancona CA. Pelvic floor muscle training in the treatment of lower urinary tract dysfunction in women with multiple sclerosis. Neurourol Urodyn. 2010 Nov;29(8):1410-3. doi: 10.1002/nau.20941. PMID 20976816
- [Background] De Ridder D, Vermeulen C, Ketelaer P, Van Poppel H, Baert L. Pelvic floor rehabilitation in multiple sclerosis. Acta Neurol Belg. 1999 Mar;99(1):61-4. PMID 10218095
- [Background] Litwiller SE, Frohman EM, Zimmern PE. Multiple sclerosis and the urologist. J Urol. 1999 Mar;161(3):743-57. PMID 10022678
- [Derived] Perez DC, Chao CW, Jimenez LL, Fernandez IM, de la Llave Rincon AI. Pelvic floor muscle training adapted for urinary incontinence in multiple sclerosis: a randomized clinical trial. Int Urogynecol J. 2020 Feb;31(2):267-275. doi: 10.1007/s00192-019-03993-y. Epub 2019 Jun 10. PMID 31183535